CLINICAL TRIAL: NCT04103333
Title: A Study to Explore Cerebrospinal Fluid and Blood Biomarkers in Participants With Angelman Syndrome
Brief Title: Angelman Syndrome (AS) Biomarker Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 992AN001
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Angelman Syndrome; Chromosome 15q Duplication (dup15q) Syndrome
MeSH Terms: conditions — Angelman Syndrome; Chromosome 15q, trisomy; Polyposis Syndrome, Hereditary Mixed, 1; Syndrome | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Angelman Syndrome: Group 1 (Experimental): Participants aged 0-6 years old with Angelman Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Angelman Syndrome: Group 2 (Experimental): Participants aged 7-12 years old with Angelman Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Angelman Syndrome: Group 3 (Experimental): Participants aged 13-18 years old with Angelman Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Angelman Syndrome: Group 4 (Experimental): Participants aged 19-50 years old with Angelman Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Dup15q Syndrome: Group 1 (Experimental): Participants aged 0-6 years old with Dup15q Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Dup15q Syndrome: Group 2 (Experimental): Participants aged 7-12 years old with Dup15q Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Dup15q Syndrome: Group 3 (Experimental): Participants aged 13-18 years old with Dup15q Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection
- Dup15q Syndrome: Group 4 (Experimental): Participants aged 19-50 years old with Dup15q Syndrome will undergo lumbar puncture (LP) for CSF and blood collection while under general anesthesia or conscious sedation during or after a prescheduled procedure unrelated to the study.
  Interventions: Procedure: Lumbar Puncture; Procedure: Blood Collection

INTERVENTIONS:
Procedure: Lumbar Puncture — Administered as specified in the treatment arm.
Procedure: Blood Collection — Administered as specified in the treatment arm.

SUMMARY:
The primary objective of this study is to measure ubiquitin-protein ligase E3A (UBE3A) protein levels in cerebrospinal fluid (CSF) and to evaluate its utility as a biomarker in support of the development of therapies for AS.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the participant's legally authorized representative (LAR) to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with national and local privacy regulations
* Must have genetically confirmed diagnosis of AS (UBE3A deletion, UBE3A mutation, paternal uniparental disomy, or imprinting center defect) or dup15q syndrome (with number and size of duplications of 15q specified) provided by the Investigator
* Must be scheduled for a procedure unrelated to the study that will involve administration of general anesthesia or conscious sedation.

Key Exclusion Criteria:

* Lumbar Puncture (LP) procedure less than 30 days before the Sampling Visit
* Any contraindications to having an LP
* The blood and CSF collection will, in the opinion of the Investigator, inhibit, in some way, the prescheduled procedure that requires anesthesia or sedation
* Current enrollment or past enrollment in an interventional clinical study in which an investigational gene therapy or antisense oligonucleotide (ASO) is/was administered
* Enrollment in an interventional clinical study in which an investigational small molecule/antibody treatment or approved small molecule/antibody therapy is administered within 1 month (or 5 half-lives of study agent, whichever is longer) prior to the Sampling Visit which, under the judgement of the Investigator and/or Sponsor would affect UBE3A and other CSF biomarker levels. Use of approved or investigational small molecule therapies which would not impact the biomarkers above will be eligible with Sponsor approval prior to enrollment (e.g., anti-epileptic drugs being studied in alternative formulation, other derivatives of benzodiazepines, or other same class drugs as those already permitted as part of the study).

Note: Other protocol defined inclusion/exclusion criteria may apply.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Ubiquitin-Protein Ligase E3A (UBE3A) Protein Levels in Each Age Group | Baseline up to Day 33
UBE3A Protein Levels in Each Genotype Group | Baseline up to Day 33

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (5):
- United States (5):
  - Rady Childrens Hospital, San Diego, California
  - Rush Medical College, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of North Carolina Hospital, Carolina, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/